CLINICAL TRIAL: NCT03751033
Title: Influence of DisCoVisc OVD on Intraoperative Aberrometry Readings for Intraocular Lens (IOL) Calculations After Cataract Extraction
Brief Title: Influence of DisCoVisc Ophthalmic Viscosurgical Device (OVD) on Intraoperative Aberrometry Readings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Consultants, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AVC-001
Record Dates: First submitted 2018-10-24; First posted 2018-11-23 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Cataract
Keywords: Cataract Extraction
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BSS and DisCoVisc (Experimental): Following lens removal and removal of all OVD from the anterior chamber during cataract surgery, the chamber will be filled with BSS and the main incision hydrated with BSS. Intraoperative aberrometry, using the Optiwave® Refractive Analysis with VerifEye+ (ORA), will be performed, and the results of aphakic refraction and suggested IOL power will be recorded in triplicate. Immediately following, the BSS will be replaced with DisCoVisc; and, triplicate readings will be measured under the same conditions.
  Interventions: Device: BSS; Device: DiscoVisc

INTERVENTIONS:
Device: BSS — Intraoperative aberrometry measurements for BSS will be performed.
Device: DiscoVisc — Intraoperative aberrometry measurements for DiscoVisc will be performed.

SUMMARY:
The purpose of the study is to develop a nomogram that correlates intraoperative, aphakic refraction measurements when the anterior chamber is pressurized with either balanced salt solution (BSS) or DisCoVisc; and to understand how suggested IOL power selection may differ.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Between 22 and 95 years of age and diagnosed with cataract(s)
* Able to comprehend and sign a written statement of informed consent for participation in the study, including HIPAA
* Undergoing cataract extraction surgery with an Alcon SN6 platform intraocular lens implantation into the posterior chamber
* Clear intraocular media, other than cataract
* Potential postoperative best-corrected visual acuity (BSCVA) of 20/30 or better
* Axial length of ≥ 22.00 and ≤ 28.00

Exclusion Criteria:

* Concurrent participation in another investigational drug or device study or participation in another study within the last 30 days prior to Screening
* Has had prior laser vision correction and/or corneal surgery
* Has a complication during surgery unrelated to ORA use
* Conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration, including pseudoexfoliation, trauma or posterior capsule defects
* History of infectious corneal disease (e.g., herpes simplex, herpes zoster, etc.) or other conditions which may result in corneal scarring
* Significant central opacity/scar
* Irregular astigmatism based upon investigator judgment
* Inability to achieve keratometric stability
* Will require another procedure, such as iris hooks, use of a Malyugin ring or insertion of a capsular tension ring during surgery
* Will require significant sedation during surgery
* Subject who is unable to maintain adequate fixation for image capture with ORA
* Keratopathy/Kerectasia - any corneal abnormality, other than regular corneal astigmatism, including, but not limited to the following: corneal leukoma and pterygium
* Any inflammation or edema (swelling) of the cornea, including but not limited to the following: keratitis, keratoconjunctivitis, and keratouveitis
* May reasonably be expected to require a secondary surgical intervention at any time during the study (other than YAG capsulotomy)
* Amblyopia
* Corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy)
* Endothelial disease that may potentially affect visual outcome
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders) that are predicted (by subjective assessment of the retina) to cause future acuity losses to a level worse than 20/30 and/or that the investigator deems would interfere with acquiring images or determining a precise postoperative refraction
* Shallow anterior chamber, not due to swollen cataract
* History of retinal detachment or macular pucker
* Ocular conditions such as keratoconus, forme fruste keratoconus or recurrent erosion syndrome that may predispose the subject to complications
* Microphthalmos
* Previous corneal transplant
* Recurrent severe anterior or posterior segment inflammation of unknown etiology
* Rubella or traumatic cataract
* Iris neovascularization
* Uncontrolled glaucoma or glaucoma with visual field defects
* Poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally
* Ectopic pupil
* Pupil abnormalities (nonreactive, fixed pupils; abnormally shaped pupils)
* Prior, current, or anticipated use during the course of the study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) likely, in the opinion of the Investigator, to cause poor dilation or lack of adequate iris structure to perform standard cataract surgery
* Aniridia
* Optic nerve atrophy
* Uncontrolled systemic disease or acute or chronic disease or illness that would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, multiple sclerosis, lupus, hepatitis, rheumatoid arthritis, etc.)
* Uncontrolled/poorly controlled diabetes
* Uncontrolled ocular hypertension (≥ 22 mmHg)
* Active intraocular inflammation or recurrent ocular inflammatory \ condition (e.g., recurrent or persistent iritis, iridocyclitis, posterior uveitis, etc.)
* Use of systemic or ocular medications that may affect vision
* Recent ocular trauma that is not resolved/stable or may affect visual outcomes
* Previous ocular surgery such as pterygium removal, tear duct surgery, radial keratectomy, etc.
* Pregnant women, nursing women and subjects suspected of being pregnant
* Subjects who, in the judgment of the investigator or sub-investigator, are inadequate for the study

Ages: 22 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Differences in aphakic refractive measurements with BSS versus DiscoVisc | 1 Day
  The differences in spherical equivalents will be evaluated using a nonparametric approach (Friedman chi-square test).

SECONDARY OUTCOMES:
Difference between suggested IOL power selections with BSS versus DiscoVisc | 1 Day
  The differences in IOL power will be evaluated using a nonparametric approach (Friedman chi-square test).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Fram, MD, Principal Investigator — Advanced Vision Care
Locations (3):
- United States (3):
  - Advanced Vision Care, Los Angeles, California
  - Cleveland Eye Clinic, Brecksville, Ohio
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No